CLINICAL TRIAL: NCT05930717
Title: Zhejiang Nutrition and Health Study: Nutrition and Lifespan Study (NuLife Study)
Brief Title: Zhejiang Nutrition and Health Study
Acronym: NuLife
Status: Withdrawn | Type: Observational
Why Stopped: The research has been withdrawn due to funding limitations.
Sponsor: Westlake University (Other)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20230511JZS001
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Disease; Cardiovascular Diseases; Healthy Aging
Keywords: Nutrition; Health; Healthy lifespan
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bio-samples mainly fasting blood, stool and urine samples will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project aims to explore the relationship between healthy lifespan and nutrition through a 10-year longitudinal study in Zhejiang Province. The cohort will include individuals in a wide range of age groups. The demographic, diet, lifestyle information, health status, and corresponding bio-samples will be collected carefully. It will give a deeper insight to the relation between nutrition and healthy aging and longevity. Ultimately, this research will contribute to evidence-based nutrition interventions to improve health outcomes and enhance quality of life.

DETAILED DESCRIPTION:
This project aims to elucidate the relationship between healthy lifespan and nutrition through the establishment of a large-scale cohort of participants and longitudinal follow-ups spanning around 10 years in Zhejiang Province. The cohort will comprise individuals in a wide range of age groups starting at 6 years old. The participants will provide demographic information, anthropometry measurements, detailed diet, lifestyle data and health status, including 3-day dietary records and long-term food intake frequency recalls. Integrated with previous information, diverse bio-samples will also be collected to establish a multi-dimensional biobank. It will give a deeper insight to the relation between nutrition and healthy aging and longevity. Ultimately, this research will contribute to the development of evidence-based nutrition designed to improve health outcomes and enhance the quality of life for individuals of all ages.

ELIGIBILITY:
Inclusion Criteria:

* Chinese citizens who have resided in the surveyed area for at least 6 months before the survey within the last 12 months.
* Aged 6 years or older.
* They are included as resident households, which are comprised of people living together in one place based on family relationships, and at least one resident with permanent household registration.

Exclusion Criteria:

* Residents living in functional zones such as construction worker dormitories, military barracks, schools, nursing homes, etc.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Permanent residents in Zhejiang Province
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2033-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of cardio-metabolic diseases | up to 10 years
  The investigators will track for occurrence of cardio-metabolic diseases by follow-up surveys collected by the Zhejiang Center for Disease Control and Prevention.

SECONDARY OUTCOMES:
Changes in fasting blood glucose | Every other year， up to 10 years
  Fasting glucose will be examined in mmol/L.
Changes in fasting blood HbA1c | Every other year， up to 10 years
  Fasting blood HbA1c will be examined in %
Changes in fasting lipid metabolism | Every other year， up to 10 years
  Triglyceride, cholesterol, high density lipoprotein cholesterol and low density lipoprotein cholesterol will be examined in mmol/L.
Changes in fasting blood highly sensitive C-reactive protein (CRP) | Every other year， up to 10 years
  CRP will be examined in mg/L.
Changes in body mass index | Every other year， up to 10 years
  Body mass index (BMI) will be calculated in kg/m^2
Changes in blood pressure | Every other year， up to 10 years
  Blood pressure, including systolic and diastolic blood pressure, will be measured in mmHg
Changes in gut microbiome profiling | Every other year， up to 10 years
  16S rRNA and/or shotgun metagenomic sequencing will be performed in stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (2):
- China (2):
  - Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou, Zhejiang
  - Westlake University, Hangzhou, Zhejiang